CLINICAL TRIAL: NCT05820984
Title: Impact of a Short Form of the SPIRIT Checklist for Peer Reviewers to Improve the Reporting of Protocols for Randomised Controlled Trials Published in Biomedical Journals: a Randomised Controlled Trial (SPIRIT-PR)
Brief Title: A Short SPIRIT Checklist for Peer Reviewers to Improve the Reporting Quality in Published Articles (SPIRIT-PR)
Acronym: SPIRIT-PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SPIRIT-PR 2019
Record Dates: First submitted 2023-04-19; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Adequate Reporting in Published Study Protocols of Randomized Controlled Trials

STUDY DESIGN:
Who Masked: Participant
Masking Description: Authors will be blinded to the intervention allocation. Editors will not be informed about the randomisation. To avoid potential bias, peer reviewers and authors will not be informed of the study hypothesis, design and intervention. All submitting authors and invited reviewers are routinely told that BMJ has a research programme and their article/review may be included in this research.
  Outcomes will be assessed in duplicate by blinded outcome assessors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIRIT checklist plus usual practice (Experimental): After accepting to review an article, peer reviewers will receive the automated, journal specific standard email with general information as per each journal's usual practice (e.g. where to access the manuscript, date when the peer review report is due). In addition, peer-reviewers who received a manuscript which was randomised to the experimental arm will receive an additional email including a short version of the SPIRIT checklist together with a short explanation of those items.
  Interventions: Other: SPIRIT checklist plus usual practice
- Usual practice (Other): After accepting to review an article, peer reviewers will receive the automated, journal specific standard email with general information as per each journal's usual practice.
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: SPIRIT checklist plus usual practice — Peer reviewer will be reminded of the following 10 CONSORT items (including a short description):
  Outcomes (12) Sample size (14) Recruitment (15) Allocation implementation (16 c) Blinding (17 a) Data collection methods (18 a) Data collection methods - retention (18 b) Statistical methods (20 a) Population analysed (20 c) Access to data (29)
  Arms: SPIRIT checklist plus usual practice
Other: Usual practice — Peer review as it is usual practice at the journal
  Arms: Usual practice

SUMMARY:
Transparent and accurate reporting is key, so that readers can adequately interpreting the results of a study. The aim of this project is to evaluate whether reminding peer reviewers of the most important SPIRIT reporting items (including a short explanation of those items) will result in higher adherence to SPIRIT guidelines in published protocols for RCTS. During the standard peer-review process, peer-reviewers will be randomly allocated to use either (i) a short version of the SPIRIT checklist including the ten most important and poorly reported SPIRIT items ; or (ii) no checklist. The aim is to find an intervention which improves the reporting, making it easier for readers to adequately interpret the presented articles.

DETAILED DESCRIPTION:
The full protocol is available on Open Science Framework where the study was prospectively registered: https://osf.io/z2hm9

ELIGIBILITY:
Inclusion criteria for journals:

It was planned from the beginning that this study will only be conducted at the BMJ Open as it publishes numerous protocols. Hence, no inclusion criteria for the journal were specified.

Inclusion criteria for manuscripts:

All submitted manuscripts sent out for external review that described protocols for RCTs.

Exclusion criterial for manuscripts:

We excluded (i) Manuscripts which were clearly labelled as a pilot or feasibility study (ii) Studies randomizing animals or cells (iii) Separate publications of data analysis plans

Included peer-reviewers:

-Peer reviewers that were invited following usual journal practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Completeness of reporting | Through study completion, an average of 1 year
  The primary outcome of this study will be the difference of the mean proportion of adequately reported items of the 10 most important and poorly reported SPIRIT items between the two intervention arms.

SECONDARY OUTCOMES:
Completeness of reporting | Through study completion, an average of 1 year
  Mean proportion of adequate reporting of the 10 most important and poorly reported SPIRIT items, considering each sub-item as a separate item.
Completeness of reporting | Through study completion, an average of 1 year
  Mean proportion for each of the 10 most important and poorly reported SPIRIT items separately (including also separate analysis of sub-items).
Time from assigning an academic editor until the first decision (as communicated to the author after the first round of peer-review). | Through study completion, an average of 4 months; will be assessed from routinely collected data
Proportion of articles directly rejected after the first round of peer-review | Through study completion, an average of 4 months; will be assessed from routinely collected data
Proportion of articles published | Through study completion, an average of 9 months; will be assessed from routinely collected data

OTHER OUTCOMES:
Peer reviewer comments for any reference to SPIRIT and trial reporting | Assessed from available peer-reviewer responses; on average 3 months after randomisation
  For journals where peer reviewer comments are subsequently published alongside the published article, we will examine the peer reviewer comments for any reference to SPIRIT and trial reporting.

CONTACTS AND LOCATIONS:
Locations (1):
- The BMJ Publishing Group, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish the anonymised data set together with the main publication.
Supporting Information: Study Protocol
Time Frame: The full protocol is publicly available on OSF (https://osf.io/z2hm9)

REFERENCES:
- [Derived] Speich B, Mann E, Schonenberger CM, Mellor K, Griessbach AN, Dhiman P, Gandhi P, Lohner S, Agarwal A, Odutayo A, Puebla I, Clark A, Chan AW, Schlussel MM, Ravaud P, Moher D, Briel M, Boutron I, Schroter S, Hopewell S. Reminding Peer Reviewers of Reporting Guideline Items to Improve Completeness in Published Articles: Primary Results of 2 Randomized Trials. JAMA Netw Open. 2023 Jun 1;6(6):e2317651. doi: 10.1001/jamanetworkopen.2023.17651. PMID 37294569